CLINICAL TRIAL: NCT01946425
Title: Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Quadrivalent Influenza Virus Vaccine (2013-2014 Formulation)
Brief Title: Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Quadrivalent Influenza Virus Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC51; U1111-1120-1262 (Other: WHO)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus vaccine; Fluzone® Quadrivalent Influenza Vaccine (No Preservative)
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Age 6 Months to <36 Months (Study Group 1) (Experimental): Participants at 6 months to < 36 months of age at enrollment
  Interventions: Biological: Fluzone® Quadrivalent Influenza Virus Vaccine, No Preservative
- Age 3 Years to <9 Years Group (Study Group 2) (Experimental): Participants at 3 years to < 9 years of age at enrollment
  Interventions: Biological: Fluzone® Quadrivalent Influenza Virus Vaccine, No Preservative

INTERVENTIONS:
Biological: Fluzone® Quadrivalent Influenza Virus Vaccine, No Preservative — 0.25 mL, Intramuscular (Pediatric Dose, 2013-2014 formulation)
  Other Names: Fluzone® Quadrivalent, No Preservative
  Arms: Age 6 Months to <36 Months (Study Group 1)
Biological: Fluzone® Quadrivalent Influenza Virus Vaccine, No Preservative — 0.5 mL, Intramuscular (2013-2014 formulation)
  Other Names: Fluzone® Quadrivalent, No Preservative
  Arms: Age 3 Years to <9 Years Group (Study Group 2)

SUMMARY:
The aim of this study is to evaluate the safety and immunogenicity of Fluzone® Quadrivalent vaccine in participants aged 6 months to < 9 years at enrollment, divided into 2 age strata (6 months to < 36 months and 3 years to < 9 years)

Primary Objective:

* To describe the safety of the 2013-2014 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule, in accordance with Advisory Committee on Immunization Practices (ACIP) recommendations, in children 6 months to < 9 years of age.

Observational Objectives:

* To describe the immunogenicity of the 2013-2014 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule in accordance with ACIP recommendations, in children 6 months to < 9 years of age.
* To submit sera from subjects to the Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), the Centers for Disease Control and Prevention (CDC), and the Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.

DETAILED DESCRIPTION:
Participants will be assigned to the appropriate age group (6 months to < 36 months of age or 3 years to < 9 years of age) based on the subject's age at the time of enrollment.

Solicited adverse event (AE) information will be collected for 7 days after each vaccination, unsolicited AE information will be collected from Visit 1 to Visit 2, or to Visit 3 for those subjects receiving 2 doses. Serious adverse event information will be collected from Visit 1 to Visit 2, or Visit 3 for those subjects receiving 2 doses.

Immunogenicity will be evaluated in all subjects prior to vaccination on Day 0 (Visit 1) and at Day 28 after the final vaccination using the hemagglutination inhibition technique. For each influenza vaccine strain, pre- and post-vaccination geometric mean titers will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 6 months to < 9 years of age on the day of first study vaccination (study product administration)
* Subject and parent/legally acceptable representative are willing and able to attend scheduled visits and to comply with the study procedures during the entire duration of the study
* Assent form has been signed and dated by subjects 7 to < 9 years of age, and informed consent form has been signed and dated by parent(s) or another legally acceptable representative
* For subjects 6 months to < 12 months of age, born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg (5.5 lbs.)

Exclusion Criteria:

* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone Quadrivalent vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information)
* History of serious adverse reaction to any influenza vaccine
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2 for subjects receiving 1 dose of influenza vaccine or Visit 3 for subjects receiving 2 doses of influenza vaccine
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study
* Prior vaccination with any formulation of 2013-2014 influenza vaccine
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular (IM) vaccination, at the discretion of the Investigator
* Thrombocytopenia, which may be a contraindication for IM vaccination, at the discretion of the Investigator
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine
* Personal history of Guillain-Barré syndrome
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Known seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F]). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Identified as a natural or adopted child of the Investigator or an employee with direct involvement in the proposed study

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- United States (2):
  - Bardstown, Kentucky
  - Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 16 September 2013 to 10 October 2013 at 2 clinic centers in the United States.
Pre-assignment Details: A total of 60 participants who met all of the inclusion and none of the exclusion criteria were enrolled and vaccinated in this study.
Groups:
- Age 6 Months to <36 Months Group: Participants 6 months to <36 months of age who received a 0.25 mL dose of Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation)
- Age 3 Years to <9 Years Group: Participants 3 years to <9 years of age who received a 0.5 mL dose of Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation)
Period: Overall Study
Arm/Group | Age 6 Months to <36 Months Group | Age 3 Years to <9 Years Group
Started | 30 | 30
Completed | 28 | 30
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Age 6 to <36 Months Group: Participants 6 months to <36 months of age who received a 0.25 mL dose of Fluzone® Quadrivalent Influenza Virus Vaccine (2013-2014 formulation)
- Age 3 to <9 Years Group: Participants 3 years to <9 years of age who received a 0.5 mL dose of Fluzone® Quadrivalent Influenza Virus Vaccine (2013-2014 formulation)
- Total: Total of all reporting groups
Arm/Group | Age 6 to <36 Months Group | Age 3 to <9 Years Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 1.9 (0.6) | 5.4 (1.8) | 3.7 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Geometric Mean Titers (GMTs) of Influenza Antibodies Before and Following Vaccination With the 2013-2014 Formulation of Fluzone® Quadrivalent, Influenza Vaccine
Description: Influenza virus antibodies were measured using a hemagglutination inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Geometric mean titers of antibodies against the hemagglutinin antigens were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Age 6 Months to <36 Months Group: Participants 6 months to <36 months of age that received Fluzone® Quadrivalent, Influenza Vaccine (2013-2014 formulation)
- Age 3 Years to <9 Years Group: Participants 3 years to <9 years of age that received Fluzone® Quadrivalent, Influenza Vaccine (2013-2014 formulation)
Arm/Group | Age 6 Months to <36 Months Group | Age 3 Years to <9 Years Group
Number analyzed (Participants) | 26 | 28
Titers
  A/H1N1 (pre-vaccination; N = 25, 28) | 14.1 [7.76 to 25.8] | 136 [68.4 to 271]
  A/H1N1 (post-vaccination; N = 26, 28) | 245 [132 to 455] | 1264 [930 to 1719]
  A/H3N2 (pre-vaccination; N = 25, 28) | 23.6 [12.5 to 44.8] | 215 [109 to 427]
  A/H3N2 (post-vaccination; N = 26, 28) | 484 [287 to 817] | 1103 [788 to 1544]
  B Yamagata (pre-vaccination; N = 25, 28) | 6.24 [4.94 to 7.88] | 29.0 [18.3 to 45.8]
  B Yamagata (post-vaccination; N = 26, 28) | 48.2 [26.7 to 87.1] | 162 [114 to 231]
  B Victoria (pre-vaccination; N = 25, 28) | 5.99 [4.76 to 7.54] | 13.1 [8.61 to 20.0]
  B Victoria (post-vaccination; N = 26, 28) | 24.8 [12.7 to 48.1] | 113 [72.8 to 176]

2. Secondary Outcome: Number of Participants With Seroprotection Before and Following Vaccination With the 2013-2014 Formulation of Fluzone® Quadrivalent, Influenza Vaccine
Description: Influenza virus antibodies were measured using an HAI assay. Seroprotection was defined as a titer ≥40 (1/dilution).
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Seroprotection against the hemagglutinin antigens were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Age 6 Months to <36 Months Group | Age 3 Years to <9 Years Group
Number analyzed (Participants) | 26 | 28
Participants
  A/H1N1 (pre-vaccination; N = 25, 28) | 5 | 19 [0 to 0]
  A/H1N1 (post-vaccination; N = 26, 28) | 22 | 28 [0 to 0]
  A/H3N2 (pre-vaccination; N = 25, 28) | 8 | 24 [0 to 0]
  A/H3N2 (post-vaccination; N = 26, 28) | 24 | 28 [0 to 0]
  B Yamagata (pre-vaccination; N = 25, 28) | 1 | 16 [0 to 0]
  B Yamagata (post-vaccination; N = 26, 28) | 18 | 27 [0 to 0]
  B Victoria (pre-vaccination; N = 25, 28) | 1 | 6 [0 to 0]
  B Victoria (post-vaccination; N = 26, 28) | 8 | 22 [0 to 0]

3. Secondary Outcome: Number of Participants Achieving Seroconversion Following Vaccination With the 2013-2014 Formulation of Fluzone® Quadrivalent, Influenza Vaccine
Description: Influenza virus antibodies were measured using an HAI assay. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and a ≥ 4-fold increase in post-vaccination titer.
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Seroconversion against the hemagglutinin antigens were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Age 6 Months to <36 Months Group | Age 3 Years to <9 Years Group
Number analyzed (Participants) | 26 | 28
Participants
  A/H1N1 (N = 25, 28) | 20 | 19 [0 to 0]
  A/H3N2 (N = 25, 28) | 22 | 14 [0 to 0]
  B Yamagata (N = 25, 28) | 17 | 17 [0 to 0]
  B Victoria (N = 25, 28) | 8 | 17 [0 to 0]

4. Secondary Outcome: Geometric Mean Titer Ratios (GMTRs) of Influenza Antibodies Following Vaccination With the 2013-2014 Formulation of Fluzone® Quadrivalent, Influenza Vaccine
Description: Influenza virus antibodies were measured using an HAI assay. Geometric mean titer ratios are the geometric means of the individual post-vaccination/pre-vaccination titer ratios for each hemagglutinin antigen contained in the vaccine.
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Geometric mean titer ratios against the hemagglutinin antigens were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer Ratio
Arm/Group | Age 6 Months to <36 Months Group | Age 3 Years to <9 Years Group
Number analyzed (Participants) | 26 | 28
Titer Ratio
  A/H1N1 (N = 25, 28) | 13.9 [8.33 to 23.3] | 8.83 [4.95 to 15.7]
  A/H3N2 (N = 25, 28) | 15.8 [9.43 to 26.4] | 4.82 [2.99 to 7.75]
  B Yamagata (N = 25, 28) | 5.13 [3.06 to 8.61] | 4.70 [3.20 to 6.90]
  B Victoria (N = 25, 28) | 2.87 [1.72 to 4.79] | 6.17 [4.17 to 9.13]

5. Primary Outcome: Number of Participants Reporting Solicited Injection-Site or Systemic Reactions Following Vaccination With the 2013-2014 Formulation of Fluzone® Quadrivalent, Influenza Vaccine
Description: Solicited injection-site reactions (6 months to <36 months of age): Tenderness, Erythema, and Swelling. Systemic reactions: Fever (Temperature), Vomiting, Crying Abnormal, Drowsiness, Appetite loss, and Irritability. Grade 3: Tenderness, Cries if limb is moved; Erythema and Swelling, ≥50 mm; Fever, >103.1ºF; Vomiting, ≥6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal, >3 hours; Drowsiness, Sleeping most of the time; Appetite lost, Refuses ≥3 feeds/meals or refuses most feeds/meals; Irritability, Inconsolable.
  Solicited injection-site reactions (3 years to < 9 years of age): Pain, Erythema, and Swelling. Systemic Reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3: Pain, Incapacitating, unable to perform usual activities; Erythema and Swelling, ≥50 mm; Fever, ≥102.1ºF; Headache, Malaise, and Myalgia, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection-site reactions and systemic reactions were assessed using the Safety Analysis Set, which includes all participants who received at least one dose of study vaccine.
Measure: Number; unit: Participants
Groups:
- Age 3 Years to <9 Years Group: Participants 3 years to <9 years of age that received Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation)
Arm/Group | Age 6 Months to <36 Months Group | Age 3 Years to <9 Years Group
Number analyzed (Participants) | 29 | 30
Participants
  Injection-site tenderness | 20 | NA — This injection-site reaction was not solicited in this group
  Grade 3 Injection-site tenderness | 5 | NA — This injection-site reaction was not solicited in this group
  Injection-site erythema | 15 | 10
  Grade 3 Injection-site erythema | 0 | 1
  Injection-site swelling | 7 | 7
  Grade 3 Injection-site swelling | 0 | 1
  Injection-site pain | NA — This injection-site reaction was not solicited in this group. | 21
  Grade 3 Injection-site pain | NA — This injection-site reaction was not solicited in this group. | 1
  Fever | 6 | 2
  Grade 3 Fever | 0 | 0
  Vomiting | 4 | NA — This systemic reaction was not solicited in this group.
  Grade 3 Vomiting | 0 | NA — This systemic reaction was not solicited in this group.
  Crying abnormal | 10 | NA — This systemic reaction was not solicited in this group.
  Grade 3 Crying abnormal | 3 | NA — This systemic reaction was not solicited in this group.
  Drowsiness | 8 | NA — This systemic reaction was not solicited in this group.
  Grade 3 Drowsiness | 1 | NA — This systemic reaction was not solicited in this group.
  Appetite lost | 7 | NA — This systemic reaction was not solicited in this group.
  Grade 3 Appetite lost | 2 | NA — This systemic reaction was not solicited in this group.
  Irritability | 17 | NA — This systemic reaction was not solicited in this group.
  Grade 3 Irritability | 3 | NA — This systemic reaction was not solicited in this group.
  Headache | NA — This systemic reaction was not solicited in this group. | 4
  Grade 3 Headache | NA — This systemic reaction was not solicited in this group. | 1
  Malaise | NA — This systemic reaction was not solicited in this group. | 11
  Grade 3 Malaise | NA — This systemic reaction was not solicited in this group. | 0
  Myalgia | NA — This systemic reaction was not solicited in this group. | 13
  Grade 3 Myalgia | NA — This systemic reaction was not solicited in this group. | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 after final vaccination.
Groups:
- Age 6 Months to <36 Months Group: Participants 6 months to < 36 months of age that received Fluzone® Quadrivalent Influenza Vaccine (2013-2014 formulation)
- Age 3 Years to <9 Years Group: Participants age 3 years to < 9 years of age that received Fluzone® Quadrivalent Influenza Vaccine (2013-2014 formulation)
Arm/Group | Age 6 Months to <36 Months Group | Age 3 Years to <9 Years Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 21/30 | 21/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Age 6 Months to <36 Months Group (N=30) | Age 3 Years to <9 Years Group (N=30)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Injection-site tenderness (General disorders) | 20/29 (20) | 0/0 (0)
Injection-site erythema (General disorders) | 15/29 (15) | 10 (10)
Injection-site swelling (General disorders) | 7/29 (7) | 7 (7)
Fever (General disorders) | 6/29 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4/29 (4) | 0/0 (0)
Crying abnormal (Psychiatric disorders) | 10/29 (10) | 0/0 (0)
Drowsiness (Nervous system disorders) | 8/29 (8) | 0/0 (0)
Appetite lost (Metabolism and nutrition disorders) | 7/29 (7) | 0/0 (0)
Irritability (Psychiatric disorders) | 17/29 (17) | 0/0 (0)
Injection-site pain (General disorders) | 0/0 (0) | 21 (21)
Headache (Nervous system disorders) | 0/0 (0) | 4 (4)
Malaise (General disorders) | 0/0 (0) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications